CLINICAL TRIAL: NCT06797830
Title: Improving Core Strength in the Warfighter With a Novel Device
Acronym: AllCore
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Moss (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, David Moss, Principal Investigator, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMCSD.2025.0010
Record Dates: First submitted 2025-01-21; First posted 2025-01-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Core Strengthening; Posture; Low Back Pain
Keywords: AllCore
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: This is a prospective observational cohort using pre and post measurements of posture and core strength in subjects treated consistently with the AllCore360. The patients will act as their own control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort (Experimental): This is a prospective observational cohort using pre and post measurements of posture and core strength in subjects (Active Duty Members enrolled in Tactical Air Control Party Training) treated consistently with the AllCore360. The patients will act as their own control.
  Interventions: Device: AllCore

INTERVENTIONS:
Device: AllCore — AllCore360° is a novel core-strengthening machine intervention designed to target trunk muscles through gravity by means of high-intensity constant velocity rotating exercise (allcore360.com).
  AllCore360° is systematic, consistent and designed for use over time. The core is strengthened because a patient's core muscles are used in anterior, lateral, and posterior contractions sequentially during a single rotation (Palevo). The patient must resist gravity with the rotation as well as contract and fire isometrically to keep proper posture. Using proper posture, the patient must keep their back straight and neck neutral throughout the length of the intervention without relying on their lower body muscles at all (this is assisted by straps rendering the legs useless and by securing the pelvis in the chair).

SUMMARY:
Low back pain is one of the most common chief complaints amongst adult patients in the ambulatory clinic and emergency settings and poor core strength is a known underlying cause/perpetuator. Additionally, it is one of the most common reasons active-duty military personnel seek medical care (absolute 2015; absolute 2016; absolute 2017). Moreover, musculoskeletal conditions represent a common reason service members are placed on limited duty and considered medically not fit to deploy. The AllCore360° has the potential to prevent pain and injury, decrease pain as well as reduce duty, fitness and mobility restrictions in active-duty members with low back pain.

DETAILED DESCRIPTION:
Trunk control enables the body to stay upright while sitting and standing. Trunk muscles also respond to shifting weight during activity in order to keep the body balanced and to prevent falling over due to shifts in center-of-gravity. Trunk control is necessary to perform activities of daily living and to stave off low back pain to ensure servicemember optimal performance. Weakened trunk muscles are a symptom of conditions such as cerebral palsy and stroke as well as causing more common conditions such as low back pain (Karthikbabu; Emami). Military pilots with weak core muscles were associated with having significant low back pain (Yang). Chinese military recruits assigned to core muscle functional strength training intervention had half as many reports of low back pain as the control group and also reported increased lumbar endurance (Wang). After 9 weeks, military police officers given trunk training had significantly lower general musculoskeletal pain than control as well as increased trunk muscle endurance (Grani). A systematic review in 2021 concluded that core stability provides therapeutic effects in patients with nonspecific low back pain by reducing pain and disability and by improving quality of life measures (Frizziero).

AllCore360° is a novel core-strengthening machine intervention designed to target trunk muscles through gravity by means of high-intensity constant velocity rotating exercise (allcore360.com). AllCore360° is systematic, consistent and designed for use over time. The core is strengthened because a patient's core muscles are used in anterior, lateral, and posterior contractions sequentially during a single rotation (Palevo). The patient must resist gravity with the rotation as well as contract and fire isometrically to keep proper posture. Using proper posture, the patient must keep their back straight and neck neutral throughout the length of the intervention without relying on their lower body muscles at all (this is assisted by straps rendering the legs useless and by securing the pelvis in the chair). AllCore360° can be individualized so that the patient is sitting at a specific degree (0° to 90°), where lowering the degree increases the difficulty of keeping muscles activated to continuecorrect posture. Once secured to the machine, the patient spends a pre-specified number of minutes with their whole body spinning in a 360° arc at the pre-specified angle programmed into the machine, rotating clockwise, counter-clockwise, or both.

AllCore360° is a relatively new machine outside of high-performance sports and intense rehab, and as such there is little published literature evaluating it. Case reports do exist. One case report showed the impact a 14-week program of AllCore360° isometric trunk training had on a child with cerebral palsy, where upon completion the patient had improved trunk stability and motor function (Park). Another case series looked at the AllCore360°'s effect on trunk function, balance, and mobility after stroke, finding improved lateral control during standing and showing that an extended program of AllCore360° sessions is feasible and repeatable (Pilkar).

ELIGIBILITY:
**Patients must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* Healthy DoD beneficiaries at Nellis Air Force Base between the ages of 18 and 50 participating in Tactical Air Control Party Specialist (TACP) training program

Exclusion Criteria:

* Legally Authorized Representatives will not be utilized in this study.
* Current low back pain
* history of spinal surgery
* history of other serious spinal pathology (e.g. annular tears, spinal stenosis [canal or neuroforaminal], fracture, painful spinal arthritis)
* pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Posture | baseline/week 1 (visit 1), week 4 (visit 12), week 7 (visit 13)
  Providers will evaluate participants posture using the PostureScreen® mobile app. The PostureScreen® mobile app can be loaded onto an iPad or phone and used by study personnel to take photos of the subject. The software then measures postures from multiple views and produces a total of 41 with the spine data (31 without the spine data) postural measurements. These measurements are reported as anterior/lateral translations and angular displacements in a scale of inches or degrees respectively. A translation or angulation of 0 would indicate no postural displacement for that specific measure. This will be measured a total of 3 times over the course of the study.
Core Strength | visit 1 (week), visit 2 (week 1), visit 3 (week 1); visit 4 (week 2), visit 5 (week 2), visit 6 (week 2); visit 7 (week 3), visit 8 (week 3), visit 9 (week 3); visit 10 (week 4), visit 11 (week 4), visit 12 (week 4); visit 13 (week 7)
  Providers will evaluate participants core strength using sEMG measurement taken by DynaROM™ Motion EMG developed by Myovision. DynaROM™ uses sEMG to measure contractile strength in microvolts (μV) of underlying the muscles during contraction. Strength of contraction of the oblique muscles and lumbar paraspinous muscles will be measured by leads placed over these respective muscle groups. Strength on muscle contractions will be recorded every 10th of a second for the entire 10-minute session. A measurement of 0 would indicate no muscle contraction. This will be measured at every visit for a total of 13 times.

SECONDARY OUTCOMES:
Core Strength -- AllCore degree setting | visit 1 (week), visit 2 (week 1), visit 3 (week 1); visit 4 (week 2), visit 5 (week 2), visit 6 (week 2); visit 7 (week 3), visit 8 (week 3), visit 9 (week 3); visit 10 (week 4), visit 11 (week 4), visit 12 (week 4); visit 13 (week 7)
  Providers will also evaluate participants core strength by recording the AllCore degree settings of each subject at each visit. The AllCore ranges from 0° to 90° and it can be adjusted at each visit according to the subject's core strength. This will be measured at every visit for a total of 13 times.

CONTACTS AND LOCATIONS:
Locations (1):
- Mike O'Callaghan Military Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
We are unable to share data.

REFERENCES:
- [Background] Boland DM, Neufeld EV, Ruddell J, Dolezal BA, Cooper CB. Inter- and intra-rater agreement of static posture analysis using a mobile application. J Phys Ther Sci. 2016 Dec;28(12):3398-3402. doi: 10.1589/jpts.28.3398. Epub 2016 Dec 27. PMID 28174460
- [Background] Cleland CL, Hunter RF, Kee F, Cupples ME, Sallis JF, Tully MA. Validity of the global physical activity questionnaire (GPAQ) in assessing levels and change in moderate-vigorous physical activity and sedentary behaviour. BMC Public Health. 2014 Dec 10;14:1255. doi: 10.1186/1471-2458-14-1255. PMID 25492375
- [Background] Clark LL, Hu Z. Diagnoses of low back pain, active component, U.S. Armed Forces, 2010-2014. MSMR. 2015 Dec;22(12):8-11. PMID 26726722
- [Background] Armed Forces Health Surveillance Branch. Absolute and relative morbidity burdens attributable to various illnesses and injuries, active component, U.S. Armed Forces, 2015. MSMR. 2016 Apr;23(4):2-7. No abstract available. PMID 27152681
- [Background] Armed Forces Health Surveillance Branch. Absolute and relative morbidity burdens attributable to various illnesses and injuries, active component, U.S. Armed Forces, 2016. MSMR. 2017 Apr;24(4):2-8. No abstract available. PMID 28488875
- [Background] Pilkar R, Veerubhotla A, Ibironke O, Ehrenberg N. A Novel Core Strengthening Intervention for Improving Trunk Function, Balance and Mobility after Stroke. Brain Sci. 2022 May 20;12(5):668. doi: 10.3390/brainsci12050668. PMID 35625054
- [Background] Armed Forces Health Surveillance Branch. Absolute and relative morbidity burdens attributable to various illnesses and injuries, active component, U.S. Armed Forces, 2017. MSMR. 2018 May;25(5):2-9. No abstract available. PMID 29799210
- [Background] Park, Eunse and Castle, Kimberly (2021) "The effect of an isometric trunk training during spinning in a child with Cerebral Palsy: A case report," Interprofessional Journal of Healthcare and Research: Vol. 1 , Article 4.
- [Background] Palevo, Gregory et al. Physiological Responses to Allcore360º Core Training System. Journal of Exercise Physiology. April 2022. Vol 24 Num 2.
- [Background] Grani G, Rodacki CLN, Lubas H, Resende EF, Hoinatski R, Sentone RG, Orr R, Paulo AC. Can training trunk musculature influence musculoskeletal pain and physical performance in military police officers? Ergonomics. 2022 Feb;65(2):265-275. doi: 10.1080/00140139.2021.1973576. Epub 2021 Sep 8. PMID 34445935
- [Background] Frizziero A, Pellizzon G, Vittadini F, Bigliardi D, Costantino C. Efficacy of Core Stability in Non-Specific Chronic Low Back Pain. J Funct Morphol Kinesiol. 2021 Apr 22;6(2):37. doi: 10.3390/jfmk6020037. PMID 33922389
- [Background] Wang X, Song WJ, Ruan Y, Li BC, Lu C, Huang N, Fang FF, Gu W. Core muscle functional strength training for reducing the risk of low back pain in military recruits: An open-label randomized controlled trial. J Integr Med. 2022 Mar;20(2):145-152. doi: 10.1016/j.joim.2021.12.002. Epub 2021 Dec 16. PMID 34969649
- [Background] Yang Y, Liu S, Ling M, Ye C. Prevalence and Potential Risk Factors for Occupational Low Back Pain Among Male Military Pilots: A Study Based on Questionnaire and Physical Function Assessment. Front Public Health. 2022 Jan 4;9:744601. doi: 10.3389/fpubh.2021.744601. eCollection 2021. PMID 35059371
- [Background] Emami F, Yoosefinejad AK, Razeghi M. Correlations between core muscle geometry, pain intensity, functional disability and postural balance in patients with nonspecific mechanical low back pain. Med Eng Phys. 2018 Oct;60:39-46. doi: 10.1016/j.medengphy.2018.07.006. Epub 2018 Aug 1. PMID 30077486
- [Background] Karthikbabu S, Verheyden G. Relationship between trunk control, core muscle strength and balance confidence in community-dwelling patients with chronic stroke. Top Stroke Rehabil. 2021 Mar;28(2):88-95. doi: 10.1080/10749357.2020.1783896. Epub 2020 Jun 23. PMID 32574524